CLINICAL TRIAL: NCT05610761
Title: Efficacy of Core Stabilization Exercises in Women With Stress and Mixed Urinary Incontinence: Randomized Controlled Trial
Brief Title: Efficacy of Core Stabilization Exercises in Women With Stress and Mixed Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Merve Dikici Yağlı, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Incontinence Rehab, IstanbulU
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; incontinence rehabilitation; incontinence exercises; core stabilization exercises
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stabilization Exercises with Kegel Exercises (Experimental)
  Interventions: Behavioral: Core stabilization exercises with Kegel exercises
- Kegel Exercises (Active Comparator)
  Interventions: Behavioral: Kegel exercises

INTERVENTIONS:
Behavioral: Core stabilization exercises with Kegel exercises — Core stabilization exercise program consists of two phases: teaching the basic movement (contraction of the Transversus abdominis and other muscles with diaphragmatic breathing) and incremental exercises added to the basic movement. The basic movement will be studied before each exercise and then the specified exercises will be added. The physiatrist will teach the exercise program to the patients. The first 6 of the 12 exercises classified according to the degree of difficulty will be performed for 5 weeks, and the next 5 weeks will be moved to the other 6 exercises. The exercises will be performed at least 3 days a week, with 10 repetitions of each movement, and the program will last for 10 weeks. Compliance with the exercise program will be questioned over the phone, and patients will be evaluated with a follow-up form before the study, at the 10th week, and at the 20th week. In addition, the Kegel exercise program specified in the other group will be applied.
  Arms: Core Stabilization Exercises with Kegel Exercises
Behavioral: Kegel exercises — Kegel Exercises The exercise will start as 2 sets of 10 repetitions in the morning and evening, and after getting used to it, it will be increased to 3 sets of 10 repetitions per day.
  The patient, lying on his back with his knees bent, feet slightly apart from each other, will try to lift the breech, urinary tract opening and vagina on the pelvic floor by counting to 5, and should not tighten your abdominal and leg muscles, and should not hold your breath while doing this exercise.
  In this way, he will count up to 5 while contracting, then he will relax by counting to 10 (after getting used to it, the holding time will be increased to 10 seconds).
  Arms: Kegel Exercises

SUMMARY:
In our study, we aimed to evaluate the effects of core stabilization exercises added to traditional Kegel exercises on incontinence and quality of life in women with stress and stress dominant mixed urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Women between the ages of 18 - 55
2. Diagnosis of stress and stress predominant mixed urinary incontinence
3. Pelvic floor muscle strength ≥ 3
4. BMI ≤ 35 kg/m2
5. ≥ 1 complaint of urinary incontinence in the last month

Exclusion Criteria:

1. Pregnancy and postpartum first 6 weeks
2. Other types of incontinence and stress type 3 incontinence
3. Urinary tract infection
4. Pelvic organ prolapse advanced stage (Stage ≥ 2)
5. History of pelvic surgery or pelvic tumor
6. Surgical treatment for urinary incontinence
7. History of serious systemic or neurological disease (Severe cardiovascular disease, advanced COPD, CVO and/or Cancer, Parkinson's etc.)
8. Severe low back and/or pelvic pain

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Vaginal Pressure Measurement with Perineometer | Baseline (before intervention), immediately after intervention, 10 weeks after intervention
  The periometer is a manometer attached to a vaginal pressure probe that evaluates pelvic floor muscle (PTC) contraction with an objective result in cmH2O. Normal vaginal pressure value is 30-60 cm H2O.
  The probe is advanced 3-5 cm towards the vagina and the patient is asked to contract the perineal muscles. 3 separate measurements are made and a score is created by taking the average of these measurements.
Change in Incontinence Severity Index (ISI) | Baseline (before intervention), immediately after intervention, 10 weeks after intervention
  ISI is a simple questionnaire consisting of questioning the frequency and amount of urine leakage, and the score consists of multiplying the answers given to these two groups of questions. Incontinence severity according to scores; mild (score 1-2), moderate (score 3-6), severe (score 8-9), and very severe (score 12).

SECONDARY OUTCOMES:
Change in Muscle Strength Examination with Digital Palpation | Baseline (before intervention), immediately after intervention, 10 weeks after intervention
  Patients lie in the supine position, knees straight and legs abducted. The physiatrist inserts two distal phalanxes and one finger into the introitus vagina and tells the patient how to contract correctly, and is asked to hold the fingers firmly. Modified Oxford Scale is used for scoring.
  Muscle strength 0: No contraction. 1: Contraction is minimal, can hold fingers for <1 second. 2: Contraction is weak, fingers are not elevated and can hold for 1-3 seconds. 3: With the contraction, the doctor's fingers elevate up to the posterior vaginal wall, can hold for 4-6 seconds, repeat 3 times. 4: Doctor's fingers elevate the posterior vaginal wall, there is a feeling of intense pressure on the fingers, can hold for 7-9 seconds, repeat 3 times. 5: He can do strong contractions for 10 seconds, repeat ≥4 times.
Change in Pad Test (24 hours) | Baseline (before intervention), immediately after intervention, 10 weeks after intervention
  The pad test is one of the objective tests that shows the presence and degree of UI. The purpose of pad tests is to determine the amount of incontinence by measuring pad weight. In these tests, the weight of the pad is weighed before and after a certain time interval (1 hour, 24 hours or 48 hours).
  In the 24-hour pad test, the pads that the patient leaks for 24 hours are collected and weighed on a sensitive scale, using a precision scale and pads whose weight is known beforehand. The amount of urine leakage is determined by subtracting the weight of the pads used from the score. Scoring; Defined as <1 g definitely dry, 2-10 g mild moderate urinary incontinence, 10-50 g severe urinary incontinence, > 50 g very severe urinary incontinence
Change in Bladder Diary (3 days) | Baseline (before intervention), immediately after intervention, 10 weeks after intervention
  Bladder diaries provide information about parameters such as fluid intake and excretion amount of the patient, urinary incontinence and frequency of urination in 24-hour periods. The patient is given 3 forms of 24 hours. He is asked to write down the information including the quality and quantity of all the liquids he has taken for 3 days, the frequency of urination during the day and night, the frequency of urinary incontinence and the triggering event on these forms, together with the hours.
Change in Incontinence Impact Questionnaire (IIQ-7) | Baseline (before intervention), immediately after intervention, 10 weeks after intervention
  Urogenital Distress Inventory (UDI-6) and Incontinence Impact Questionnaire (IIQ-7) assess symptom distress and the impact on daily life of urinary incontinence. The patient is asked 7 different questions about how much urinary incontinence affects him in social life. Indicate the degree of being affected in 7 subjects: doing housework, aerobic activities such as walking, swimming, exercise, entertainment activities (such as movies), traveling for more than 30 minutes by car, participation in social activities outside the home, mental health (nervousness, depression), and feelings of frustration. required. 0 is not affected at all, 1 is slightly affected, 2 is moderately affected, and 3 is very affected.
Change in Urogenital Distress Inventory (UDI-6) | Baseline (before intervention), immediately after intervention, 10 weeks after intervention
  Urogenital Distress Inventory (UDI-6) and Incontinence Impact Questionnaire (IIQ-7) assess symptom distress and the impact on daily life of urinary incontinence. UDI-6 consists of 6 items: Frequent urination, leakage related to feeling of urgency, leakage related to activity, coughing, or sneezing small amounts of leakage (drops), difficulty emptying the bladder, and pain or discomfort in the lower abdominal or genital area. They are asked to score how much these items affect the quality of life. 0 is not affected at all, 1 is slightly affected, 2 is moderately affected, and 3 is very affected.
Change in King's Health Questionnaire (KHQ) | Baseline (before intervention), immediately after intervention, 10 weeks after intervention
  The King's Health Questionnaire (KHQ) is another comprehensive patient statement-based scoring used to evaluate the impact of urinary incontinence on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Dikici Yağlı, MD, Principal Investigator — Istanbul University; Ayşe Karan, Professor, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322